CLINICAL TRIAL: NCT03312218
Title: Can an App Improve the Examination Scores of Family Medicine Residents? A Cluster Randomized Controlled Trial
Brief Title: The Study Guide Cluster Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: Western University, Canada (Other); College of Family Physicians of Canada (Other); Memorial University of Newfoundland (Other); Université de Montréal (Other); University of Ottawa (Other); Queen's University, Kingston, Ontario (Other); University of Toronto (Other); McMaster University (Other); University of British Columbia (Other); University of Alberta (Other); Université de Sherbrooke (Other); University of Calgary (Other)
Responsible Party: Principal Investigator, Roland Grad, Associate Professor, McGill University Dept. of Family Medicine, Director of the Clinician Scholar Program, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: The Study Guide Trial 2017
Record Dates: First submitted 2017-10-06; First posted 2017-10-17 (Actual); Results first posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention site residents will receive alerts through an app to adaptively reinforce the learning of clinical content based on cases and test questions (spaced education).
  Interventions: Behavioral: Spaced educational intervention
- Control (No Intervention): Residents in the control group will receive the same app providing identical clinical cases and test questions-on-demand, but with alerts inactivated (no spaced education).

INTERVENTIONS:
Behavioral: Spaced educational intervention — A spaced educational intervention will be provided to participants
  Arms: Intervention

SUMMARY:
Spaced education is a promising theory-driven strategy to improve clinical competence. Our aim is to improve the clinical competence of Family Physicians, an outcome associated with the quality of care delivered to Canadians.

DETAILED DESCRIPTION:
Research Question: Among family medicine residents, does enhanced feedback through an app providing alerts and test questions (spaced education), compared to the same app without alerts and enhanced feedback (no spaced education), improve competence as measured by the certification examination? In building this proposal for a definitive trial, the investigators have support from coast to coast. In addition to key clinician educators, the team includes knowledge users from the organization responsible for the certification examination in Family Medicine, methodologists and experienced researchers who study how mobile apps can promote engagement with clinical information. The team has the right blend of expertise in medical education and cluster randomized trials.

Approach and Methods: The investigators will follow an organizational participatory research approach, and propose a cluster randomized controlled trial. Setting: All incoming family medicine residents in Canada will be eligible to participate. Intervention site residents will receive alerts through an app to adaptively reinforce the learning of clinical content based on cases and test questions (spaced education). Residents in the control group will receive the same app providing identical clinical cases and test questions-on-demand, but with alerts inactivated (no spaced education). The primary outcome will be scores on the certification examination. This routinely collected data will be provided to the team by the College of Family Physicians of Canada.

Expected Results and Conclusion: Spaced education will improve examination scores. This will inform educational practice by providing evidence to optimize the training of residents.

ELIGIBILITY:
Inclusion Criteria:

* incoming family medicine residents in Canada (July 2017)

Exclusion Criteria:

* not a family medicine resident
* did not start residency on July 1, 2017

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 335 | 299
Completed | 281 | 241
Not Completed | 54 | 58
Not completed — Never signed in to access the app | 54 | 58

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 335 | 299 | 634
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 335 | 299 | 634
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Disclosed gender (included 6 undisclosed in male intervention count): Female | 229 | 210 | 439
  Disclosed gender (included 6 undisclosed in male intervention count): Male | 106 | 89 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 335 | 299 | 634
Region of Enrollment [Number; unit: participants]
  Canada | 335 | 299 | 634
Smart phone [Count of Participants; unit: Participants] | 234 | 213 | 447
International Medical Graduate [Count of Participants; unit: Participants] | 40 | 57 | 97
Graduate degree [Count of Participants; unit: Participants] | 80 | 66 | 146

OUTCOME MEASURES:

1. Primary Outcome: Scores on the Certification Examination
Description: This is the score on the written component of the examination of the College of Family Physicians of Canada. This refers to the grade/score given to participants on the Short Answer Management Problems (SAMP) section of the exam ranging from 0 to 100. Higher values represent a better outcome. The score minimum observed was 53.9 and max is 84.4 for this study.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 281 | 241
scores on a scale | 73.9 (4.4) | 73.1 (5.1)

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed.
Description: Adverse Events were not monitored/assessed. The meaning of "0" Total Number of Participants at Risk is stated because adverse events were not monitored.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03312218/Prot_SAP_000.pdf